CLINICAL TRIAL: NCT05867238
Title: Impact of Stress Management Training on the Resilience and Stress of Student Nurse Anaesthetists
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 00010254 - 2023 - 033
Record Dates: First submitted 2023-05-05; First posted 2023-05-19 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Stress, Psychological
Keywords: Resilience; Acute stress; sleep quality; Anaesthetist; chronic stress
MeSH Terms: conditions — Stress, Psychological; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Student nurse anaesthetists with no training in stress management: Student nurse anaesthetists who participated in the previous study: stress of anaesthesia professionals in the operating theatre and did not receive stress management training.
- Student nurse anaesthetists with training in stress management: Volunteer nurse anaesthetist students who have received training in stress management this year.
  Interventions: Other: Training stress management

INTERVENTIONS:
Other: Training stress management — The stress management training included 1 day and a half day. It was given by a therapist trained in transactional analysis and a trainer from the nurse anaesthetist school. The training was based on cognitive behavioural stress management training and the use of stress management exercises: cardiac coherence, mindfulness meditation, muscle relaxation, mental imagery.
  Groups: Student nurse anaesthetists with training in stress management

SUMMARY:
The study aims to evaluate the effectiveness of stress management training provided to student nurse anaesthetists on: their level of chronic perceived stress in the last month, their level of acute perceived stress each day for one month, their level of resilience and their level of sleep quality.

DETAILED DESCRIPTION:
This trial will be conducted at the CHU Grenoble Alpes (CHUGA). Volunteer nurse student anaesthetists trained in stress management will complete questionnaires assessing resilience, perceived stress over the past month, sleep quality and will assess perceived stress on each working day using the visual analogue stress scale over 3 periods of the working day.

The results of the trained students will be compared to the results of the untrained students who participated in the Anaesthesia worker stress in the Operating Room survey registered under the clinical trial number: NCT05392972

The main objective is to evaluate the impact of stress management training provided to nurse anaesthetist students on their chronic perceived stress over one month assessed with the Perceived Stress Scale 10.

The secondary objectives are:

1. To compare the level of resilience of students who have received training in stress management methods with that of students who have not received such training. (Comparison of the average of the Connor-Davidson resilience scale for each population)
2. Compare the perceived stress during a working day in students who have received stress management training to those who have not. (Comparison of the average of the two visual analogue stress scales (VAS Stress) (start of shift/end of shift) collected on working days over a period of one month for both populations)
3. Compare the stress peaks experienced (acute stress) by students who have received stress management training and those experienced by students who have not. (Comparison of the median of the stress VAS peaks of the two populations followed over one month).
4. Determine whether the quality of sleep of the students is influenced by the stress management training (comparison of the pittsburgh sleep quality index (PSQI) of the nurse student anaesthesist population that received stress management training with the PSQI of population that did not receive this training).
5. Conduct a satisfaction survey among the nurse student anaesthesist regarding the training provided by the Grenoble training institute and identify the stress management methods retained as useful by the nurse student anesthesist following this training.

ELIGIBILITY:
Inclusion Criteria:

* Student nurse anaesthetist

Exclusion Criteria:

* Student objecting to the use of their personal information
* Student on study leave.
* Student on sick leave during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Student nurse anaesthetist from the Grenoble school.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale 10 | at day 30
  The Perceived Stress Scale (PSS10 from 10 To 50) measures the degree to which respondents feel their lives are unpredictable, uncontrollable, and overloaded. A high score indicates more stress.

SECONDARY OUTCOMES:
Resilience | at Day 0
  Measurement of resilience by Connor-Davidson Resilience Scale 10 (CDRISC10 from 0 to 40) in participants. A high score indicates better resilience.
Self-reported stress at the beginning of the workday. | Each work day at the start of the shift. From day 0 to day 30.
  Stress level self reported by participants on visual analogical scale (VAS from 0 to 100); One end of the scale represents the maximum conceivable symptom strength (i. e., 100%), the other end no symptoms whatsoever (i. e., 0%).
Self-reported stress at the end of the workday. | Every working day at the end of the shift. From day 0 to day 30.
  Stress level self reported by participants on visual analogical scale (VAS from 0 to 100); One end of the scale represents the maximum conceivable symptom strength (i. e., 100%), the other end no symptoms whatsoever (i. e., 0%).
Maximum self-reported stress of the workday. | Every working day at the end of the shift. From day 0 to day 30.
  Stress level self reported by participants on visual analogical scale (VAS from 0 to 100); One end of the scale represents the maximum conceivable symptom strength (i. e., 100%), the other end no symptoms whatsoever (i. e., 0%).
The score of the Pittsburgh Sleep Quality Index (PSQI) | at day 30
  The PSQI contains 19 self-assessed questions. These 19 questions combine to yield 7 components: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) habitual sleep efficiency, (5) sleep disturbance, (6) use of sleeping medication, and (7) daytime dysfunction. Each component gives a score from 0 to 3 points (0 indicates no difficulty, while 3 indicates major difficulty). The scores of the seven components are then added together to give an overall score of 0 to 21 points (0 indicating no difficulty, and 21 indicating major difficulty).
overall satisfaction with the stress management training received | at day 30
  Scale from 0 to 10 or a higher score indicates a higher level of satisfaction.
Have you implemented any of the stress management methods proposed during the training? | at day 30
  Yes or No (qualitative)
What method of stress management is used? | at day 30
  choice among: cardiac coherence,self-hypnosis,mental imagery (colourful garden),muscle relaxation,automatic thinking (safe place),rational thinking (autogenic training),breathing meditation, other / free response
If you used stress management methods: how frequently? | at day 30
  choice among : Daily,Weekly,Monthly,The day before an exam,During training periods

CONTACTS AND LOCATIONS:
Overall Officials: Julien Picard, Principal Investigator — University Hospital, Grenoble; Yoann Zafiriou, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Grenoble Hospital, Grenoble, France